CLINICAL TRIAL: NCT05329870
Title: Does Genetic Susceptibility for Bleeding Affect Quantitative Faecal Immunochemical Test (qFIT) Results? - a Feasibility Study
Brief Title: Does Genetic Susceptibility for Bleeding Affect Quantitative Faecal Immunochemical Test (qFIT) Results?
Status: Withdrawn | Type: Observational
Why Stopped: never started due to funding/staffing issues
Sponsor: University of Edinburgh (Other)
Collaborators: Royal College of Surgeons of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC21145
Record Dates: First submitted 2022-01-05; First posted 2022-04-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer; Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA will be collected and stored in the IGC Unit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Colonoscopy and Normal qFIT: Normal colonoscopy and qFIT <10 micrograms haemoglobin
  Interventions: Other: SNP array
- Normal Colonoscopy and Raised qFIT: Normal colonoscopy and qFIT >=10 micrograms haemoglobin
  Interventions: Other: SNP array

INTERVENTIONS:
Other: SNP array — SNP arrays for known bleeding SNPs to compare genetics of patients with normal colonoscopy and normal qFIT vs raised qFIT

SUMMARY:
Quantitative faecal immunochemical testing (qFIT) is used to test for blood within faeces that cannot always be visible. The presence of blood in the stool has been shown to be a finding where there may be a problem within the large bowel. The test is able to give a numeric value to the blood in the stool and based on this result, further investigations can be planned, or if normal reassurance given.

The test is not perfect and minor bowel problems such as haemorrhoids (piles) can give a raised result. However, we have also seen raised results in people who when investigated have a completely normal large bowel. A small degree of 'physiological' non-visible bleeding is likely a normal part of life and for the majority this does not lead to a raised qFIT result.

It may be the case in people who have a raised qFIT but then go on to have a completely normal colonoscopy (telescope investigation of the large bowel) that there is a genetic predisposition that increases the amount of normal 'physiological blood' that they produce. This leads to the test being falsely positive and the person undergoing an unnecessary investigation.

This study aims to use saliva to test for known genetic markers that effect blood clotting and can increase how much someone bleeds. By comparing the occurrence of these genetic markers in people with a raised qFIT and normal colonoscopy to those with a normal qFIT and normal colonoscopy, we can test this theory. Should this be the case it will help explain why the test can be raised in normal large bowel and could lead to different levels of positivity being used for different people.

DETAILED DESCRIPTION:
Quantitative faecal immunochemical testing (qFIT) measures the presence of haemoglobin within faeces. It is an immunoassay based method, measuring the globin portion of human haemoglobin or its early degradation products. Diet does not impact the result and because globin is broken down by gastric enzymes, it is more specific to lower gastrointestinal (GI) bleeding than previously used guaiac based occult blood tests. qFIT is the test currently used by the Scottish and English National Bowel Screening Programmes and more recently has been included in NICE guideline DG30, for the investigation of patients with lower gastrointestinal (GI) symptoms who are in a low-risk population.

qFIT is being increasingly used in a manner, unsupported by evidence in some cases, in the investigation of all symptomatic patients to aid decision-making in referral to secondary care and for allocation of endoscopy resources in secondary care. qFIT is not a perfect test to rule out colorectal cancer, a meta-analysis within a symptomatic population estimated the sensitivity for detecting colorectal cancer to be 90% with a specificity of 87%. From our own studies of repeated qFIT (n=3000, unpublished), a large variance is seen between the results. Therefore to improve the utility of qFIT within this group it is likely additional factors will also need to be considered, such as an individual's genetic susceptibility for bleeding.

There are well known genetic variants resulting in coagulopathy conditions such as haemophilia and von Willebrand disease. However, it has been shown that the levels of coagulation associated proteins vary within the population and this variation is linked with genetics. Multiple genes have been implicated in coagulation, and within them hundreds of singe nucleotide polymorphisms (SNPs). Reduced levels of circulating coagulation proteins may explain false positive cases seen with qFIT.

This study aims to add further knowledge to the utility of qFIT when investigating patients with lower gastrointestinal symptoms. There are a significant proportion of people who have a raised qFIT and normal colonoscopy (gold standard investigation). In our data approximately 10% of those with a completely normal colonoscopy had a raised qFIT defined as >10 µg Hb/g. It is possible that these patients have a genetic susceptibility to bleeding and therefore have higher levels of faecal haemoglobin without any pathology. There are known genetic markers for bleeding tendency. By comparing these genetic traits in patients with a normal colonoscopy but a qFIT >10 µg Hb/g against <10 µg Hb/g the potential effects of these genes on qFIT results may be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were symptomatic at the time of referral
* Returned at least one qFIT sample
* Underwent a complete colonoscopy, which did not identify any pathology
* Willing to provide a saliva sample for genetic analysis
* Are able to consent to the study

Exclusion Criteria:

* Age < 18
* Previous colorectal cancer
* Ongoing colonic polyp surveillance
* Known inflammatory bowel disease
* Taking anticoagulant medication (Aspirin, clopidogrel, warfarin or NOAC)
* History of liver disease or known bleeding disorder
* Incomplete colonoscopy
* Unable to consent to the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study would aim to enrol 150 participants. This would be in a 1:4 ratio, meaning 30 participants would have had a normal colonoscopy and a qFIT >10 µg Hb/g and 120 participants would have a normal colonoscopy and a qFIT <10 µg Hb/g.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-18 (Estimated); Primary Completion 2023-11-04 (Estimated); Study Completion 2023-11-04 (Estimated)

PRIMARY OUTCOMES:
Accumulation of SNPs related to bleeding in patients with a normal colonoscopy and a raised qFIT compared to those with a qFIT less than 10 µg Hb/g. | Saliva sample will be collected within 1 month of recruitment. Assessment will require all results from the study participants before analysis can be performed. Aimed to be within 6 months of sample collection completion
  SNP array performed on dna from saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Farhat Din, FRCSed, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pseudo-anonymised genetic profiles may be available with patient consent